CLINICAL TRIAL: NCT06067048
Title: Phase II Trial of Zanubrutinib in Primary Cold Agglutinin Disease. CaZa Study
Brief Title: Zanubrutinib in Primary Cold Agglutinin Disease
Acronym: HOVON169CAD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO169
Record Dates: First submitted 2023-07-12; First posted 2023-10-04 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Zanubrutinib, 320 mg per day (four 80 mg capsules)
  Interventions: Drug: Zanubrutinib Oral Capsule

INTERVENTIONS:
Drug: Zanubrutinib Oral Capsule — 36 cycles (1 cycle is 28 days)
  Other Names: Brukinsa

SUMMARY:
Cold agglutinin disease (CAD) is defined as a chronic autoimmune hemolytic anemia (AIHA) with a monospecific direct antiglobulin test (DAT) strongly positive for C3d and the presence of cold agglutinins (CA; titer ≥ 64 at 4°C). Patients may have a B-cell clonal lymphoproliferative disorder (LPD) detectable in blood or marrow but no clinical or radiological evidence of malignancy. CAD can lead to AIHA, peripheral ischemic symptoms (cold-induced peripheral symptoms such as acrocyanosis etc.), or both. The CAs are typically monoclonal IgM antibodies produced by the clonal B-cells, usually IgM kappa with specificity for the I antigen on erythrocytes. There is no curative treatment. Current treatment options include rituximab monotherapy, however this has only a limited and short-lasting effect. Rituximab in combination with chemotherapy induces deeper and more durable responses, however since CAD patients typically do not have an overt malignancy this comes with concerns about short- and long-term toxicity. Novel complement inhibitors may be effective for the hemolysis but are not expected to be effective against cold induced peripheral symptoms while this is directly IgM mediated. Bruton Tyrosine Kinase inhibitors (BTKis) are effective in many B-cell lymphoproliferative disorders including the IgM producing clone of Waldenström macroglobulinemia (WM) and were very effective on both AIHA and peripheral ischemic symptoms in patients with CAD based on retrospective data.

ELIGIBILITY:
INCLUSION criteria

In order to be eligible to participate in this study, a patient must meet all of the following criteria:

CAD diagnosis defined by the combination of:

1. Chronic hemolysis (>3 months; suppressed haptoglobin) and
2. Cold agglutinin titer of 64 or higher at 4°C and
3. Positive direct antiglobulin test, strongly positive (at least 2+) with anti-C3d and negative or weakly positive (maximum 2+) with anti-IgG,

AND:

The presence of a clonal B-cell lymphoproliferative disorder defined by:

1. M-protein by serum electrophoresis confirmed by immunofixation, and/or
2. A clonal CD20 positive lymphocyte population in the bone marrow (a very small clone visible only by flow cytometry is allowed)

Indication for therapy:

Hb ≤ 10.5 g/dL

AND/OR

Considerable CIPS (grade 2 or more; see appendix E)

Relapsed or refractory after at least one prior CAD treatment, OR is treatment naïve and not eligible for currently available treatment options, per clinician's judgement.

Age ≥ 18 years.

ECOG/WHO performance status ≤ 2 (see appendix B). WHO performance status 3 is allowed if related to the CAD.

Adequate bone marrow function as defined by:

Absolute neutrophil count (ANC) > 1.0 × 109/L, and

Platelets ≥ 100 x109/L.

Ferritin levels above the lower limit of normal (LLN). Concurrent treatment with iron supplementation is permitted if the patient has been on a stable dose during the previous 4 weeks.

Total bilirubin level above the upper limit of normal (ULN), as a measurable parameter for hemolysis, and that is not attributable to Gilbert's syndrome.

Negative pregnancy test at study entry for woman of childbearing potential.

Women of childbearing potential must be: (1) surgically sterile or ≥ 2 years after the onset of menopause; (2) willing to use a highly effective contraceptive method such as oral contraceptives, intrauterine device, or sexual abstinence during study treatment and for ≥ 90 days after last dose of zanubrutinib.

Male patients with a female partner of childbearing potential are eligible if vasectomized or if they agree to the use of barrier contraception with other methods as described above during the study treatment period and for ≥ 90 days after the last dose of zanubrutinib.

Written informed consent.

Patient is capable of giving informed consent and can understand and agrees to comply with the requirements of the study and the schedule.

EXCLUSION criteria ( see below)

A patient who meets any of the following criteria cannot be included in this study:

A diagnosis of agressive lymphoma, chronic lymphocytic leukemia (CLL), or the presence of overt extramedullary B-cell lymphoproliferative disease. (Note: presence of a B-cell lymphoproliferative disorder, limited to the bone marrow, including WM, MZL or IgM MGUS, is allowed. However, the indication for treatment should be only cold agglutinin-related, as per inclusion criteria.)

Cold agglutinin syndrome (CAS) secondary to specific infection (Mycoplasma or Epstein-Barr virus) or rheumatological disorders

Mixed AIHA, Evans syndrome (concurrent autoimmune thrombocytopenia/ITP).

Prior non-lymphatic malignant disease within the past 3 years, except for curatively treated basal or squamous cell skin cancer, non-muscle-invasive bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score 6 prostate cancer.

History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of unexplained spontaneous bleeding requiring blood transfusion or other medical intervention.

History of stroke or intracranial hemorrhage within 6 months before first dose of study drug.

Previous treatment with BTKi.

Major surgery within 4 weeks of the first dose of study drug.

Requiring ongoing treatment with warfarin or warfarin derivatives. Please note: Patients being treated with DOACs (e.g., apixaban, edoxaban or rivaroxaban) or antiplatelet therapy can be included, but must be properly informed about the increased risk of hemorrhage under treatment with zanubrutinib.

Requiring ongoing treatment with a moderate or strong CYP3A inducer. Patients requiring ongoing treatment with a CYP3A inhibitor (see Appendix G) can be included (with an adjusted dose of zanubrutinib).

Requiring ongoing treatment with systemic corticosteroids for an indication other than AIHA/CAD at a dose of > 10 mg prednisone per day.

Previous CAD treatment within the following time frames:

rituximab, or bortezomib monotherapy within 3 months prior to inclusion

bendamustine, fludarabine or other cytotoxic therapy with or without rituximab, or bortezomib with rituximab, within 4 months prior to inclusion

anticomplement therapies within 5 half-lives of the specific drug prior to inclusion

Erythropoietin use, which has not been at a stable dose within 3 months prior to inclusion

Clinically significant cardiovascular disease including one of the following:

1. Myocardial infarction within 6 months before screening
2. Unstable angina within 3 months before screening
3. New York Heart Association (NYHA) class III or IV congestive heart failure (see appendix D)

d History of clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes)

e. QTcF > 480ms based on Fridericia's formula

f. History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place

g. Uncontrolled hypertension as indicated by a minimum of 2 consecutive blood pressure measurements showing systolic blood pressure > 170 mmHg and diastolic blood pressure > 105 mmHg at screening

Severe or debilitating pulmonary disease (CTCAE grade III-IV, see appendix D).

Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.

Significant renal dysfunction (creatinine clearance < 30 mL/min after rehydration as estimated by the Cockcroft-Gault equation or the Modification of Diet in Renal Disease [MDRD] equation or as measured by nuclear medicine scan or 24-hour urine collection).

Significant hepatic dysfunction (transaminases ≥ 2.5 times ULN and/or serum direct bilirubin ≥ 2 x ULN). ( Elevated indirect (unconjugated) bilirubin is accepted if this is related to active hemolysis.

Uncontrolled HIV infection. Patients with HIV positivity but controlled infection (= sustained negative viral load) may be enrolled.

Known hepatitis B infection with serologic status: presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Patients with presence of HBcAb, but absence of HBsAg, are eligible if HBV DNA is undetectable (< 20 IU/mL), and if they are willing to undergo monitoring for HBV reactivation.

Presence of Hepatitis C (HCV) antibody.

Active fungal, bacterial and/or viral infection requiring systemic therapy.

Known active or latent mycobacterial infection.

Vaccination with a live vaccine within 28 days prior to the first dose of study drug.

Pregnant or breastfeeding women.

Current participation in another interventional clinical trial.

Underlying medical conditions that, in the investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of toxicity or AEs, including

severe neurological, psychological, familial, sociological or geographical condition which would compromise ability to comply with study procedures, or is accompanied by a life expectancy of < 6 months.

History of intolerance to the active ingredients or other ingredients of zanubrutinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
CAD response rate (PR or CR) after 6 cycles of zanubrutinib treatment | 1 year

SECONDARY OUTCOMES:
Rate of CAD response categories (CR, PR or none; separately) after 6 cycles of treatment and best CAD response on protocol | 3 years
Time to CAD response and time to best CAD response. | 3 years
Hematological response rates after 6 cycles, as per the classification criteria defined by the IWWM-6. | 3 years
Best hematological response rates on protocol, as per the classification criteria defined by the IWWM-6 | 3 years
Duration of CAD response and duration of hematological response | 3 years
Change in IgM, M-protein, Hb and hemolytic parameters (bilirubin, LDH) after 6 cycles compared to baseline including median change and maximal change overall on protocol | 3 years
Percentage of patients with cold-induced symptoms at baseline that achieve improvement or resolution of these symptoms after 6 cycles and overall on protocol. | 3 years
Time for patients with cold-induced symptoms at baseline to achieve improvement or resolution of these symptoms. | 3 years
Time to transfusion independence (in patients that are transfusion dependent at baseline) | 3 years

OTHER OUTCOMES:
Progression free survival, defined as time from registration to relapse of CAD or death from any cause, whichever comes first | 3 years
Time to next CAD treatment (off protocol). | 3 years
Overall survival, defined as time from registration to death from any cause. Patients alive will be censored at the date of last contact. | 3 years
Toxicity as defined by type,frequency and severity of adverse events according to the NCI Common Terminology Criteria for Adverse Events version 5.0. | 3 years
Percentage of patients completing at least 6 cycles and percentage completing the total 36 cycles of treatment | 3 years
Relative dose intensity (DI) of zanubrutinib, based on the ratio of received zanubrutinib dose to the planned dose intensity. | 3 years
Impact of zanubrutinib treatment on CIPS measured with CIPS questionnaire | 3 years
Impact of zanubrutinib treatment on patient-reported fatigue, measured by the Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-Fatigue) | 3 years
The incidence of toxicity-related dose reduction, presented as percentages of the total study population who receive reduced doses | 3 years
The incidence of CYP3A inducer-related dose reduction, presented as percentages of the total study population who receive reduced doses due to concomitant use of CYP3A inducers. | 3 years

CONTACTS AND LOCATIONS:
Locations (10):
- Belgium (2):
  - UZ leuven, Leuven
  - AZ Delta, Roeselare
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Netherlands (3):
  - Amsterdan UMC ( location AMC), Amsterdam
  - UMCG, Groningen
  - Erasusmc, Rotterdam
- Norway (3):
  - Haukeland University Hospital Bergen, Bergen
  - Oslo University Hospital, Oslo
  - st. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: HOVON website — https://hovon.nl/en